CLINICAL TRIAL: NCT00457626
Title: An Open Label Extension Study to Evaluate Safety, Tolerability, and Efficacy of 18 Weeks of Valsartan Treatment in Children 6 Months-5 Years Old With Hypertension
Brief Title: A Study to Evaluate the Long-term Use of Valsartan in Children 6 Months to 5 Years Old With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489K2303E1; 2006-005473-21 (EudraCT Number)
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Children; pediatrics; High Blood Pressure; Hypertension; Valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valsartan Open Label (Experimental): Extemporaneous oral suspension prepared from valsartan tablets was administered to participants once daily. The starting dose of valsartan was 1 mg/kg, escalated to 2 mg/kg or 4 mg/kg based on mean sitting systolic blood pressure (MSSBP) control after 2 weeks up to 18 weeks.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — Extemporaneous suspension of valsartan, orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of long-term use (up to 18 weeks) of valsartan in children 6 months to 5 years old with hypertension.

ELIGIBILITY:
Inclusion criteria

* Participants who qualified and entered the core study.
* Participants who participated in the core study, completed Period 1 and were re-randomized in Period 2 and continued for at least 3 days in Period 2.

Exclusion criteria

* Participants who did not complete Period 1 of the core study.
* Participants who were re-randomized in Period 2 of core study but did not continue for => 3 days in Period 2 of the core study.
* Participants who experienced any adverse events considered serious or drug related in the core study.
* Participants excluded from the core study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2007-04-09 (Actual); Primary Completion 2009-05-25 (Actual); Study Completion 2009-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- United States (3):
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Norfolk, Virginia
- Belgium (5):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Recife, Pernambuco
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- India (6):
  - Novartis Investigative Site, Hyderabad, Andh Prad
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Indore, M.P.
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, New Delhi
- Italy (2):
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Palermo
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
- South Africa (4):
  - Novartis Investigative Site, Gezina, Gauteng
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Potchefstroom
  - Novartis Investigative Site, Pretoria
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir

REFERENCES:
- [Result] Schaefer F, Coppo R, Bagga A, Senguttuvan P, Schlosshauer R, Zhang Y, Kadwa M. Efficacy and safety of valsartan in hypertensive children 6 months to 5 years of age. J Hypertens. 2013 May;31(5):993-1000. doi: 10.1097/HJH.0b013e32835f5721. PMID 23511339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 investigative sites in 10 countries from 9 April 2007 to 25 March 2009.
Pre-assignment Details: This study enrolled a total of 66 participants who completed the core study (NCT00435162).
Groups:
- Valsartan Open Label: Extemporaneous oral suspension prepared from valsartan tablets was administered to participants once daily. The starting dose of valsartan was 1 mg/kg escalated to 2 mg/kg or 4 mg/kg based on mean sitting systolic blood pressure (MSSBP) control after 2 weeks up to 18 weeks.
Period: Overall Study
Arm/Group | Valsartan Open Label
Started | 66
Completed | 60
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Administrative Problems | 2
Not completed — Participant's Condition No Longer Requires Study Drug | 1

BASELINE CHARACTERISTICS:
Population: Enrolled extension participants (ENRE) included all participants who were enrolled into this extension study.
Arm/Group | Valsartan Open Label
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participant remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 1-2 minute intervals and the mean of three sitting systolic blood pressure (SSBP) measurements were used as the average sitting office blood pressure for that visit. Negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 26
Population: The extension set (ESET) included all participants who entered the extension study, with administration of at least one dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Groups:
- Valsartan Open Label: Extemporaneous oral suspension prepared from valsartan tablets was administered to participants once daily. The starting dose of valsartan was 1 mg/kg escalated to 2 mg/kg or 4 mg/kg based on MSSBP control after 2 weeks up to 18 weeks.
Arm/Group | Valsartan Open Label
Number analyzed (Participants) | 66
millimeters of mercury (mmHg)
  Baseline | 114.7 (9.04)
  Change from Baseline at Week 26 | -11.2 (12.56)

2. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participant remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 1-2 minute intervals and the mean of three SDBP measurements were used as the average sitting office blood pressure for that visit. Negative change from Baseline indicates improvement.
Time Frame: Baseline to Week 26
Population: The ESET included all participants who entered the extension study, with administration of at least one dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan Open Label
Number analyzed (Participants) | 66
mmHg
  Baseline | 70.7 (11.14)
  Change from Baseline at Week 26 | -6.6 (11.84)

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participant or require medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: Week 8 to Week 26 of Extension Phase
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Valsartan Open Label
Number analyzed (Participants) | 66
Participants
  AEs | 38
  SAEs | 4

ADVERSE EVENTS:
Time Frame: Week 8 to Week 26 of Extension Phase
Description: The ESET included all participants who entered the extension study, with administration of at least one dose of open-label study drug.
Arm/Group | Valsartan Open Label
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 4/66
Other Adverse Events (participants affected / at risk) | 38/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan Open Label (N=66)
Viral infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan Open Label (N=66)
Diarrhoea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 11
Bronchitis (Infections and infestations) | 5
Ear infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 2
Viral infection (Infections and infestations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.